CLINICAL TRIAL: NCT01141803
Title: Isafruit: Nutrigenomics in Overweight
Brief Title: Effect of Apple and Apple Pomace on Inflammation and Cholesterol Metabolism in Healthy Overweight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Technical University of Denmark (Other); Central Jutland Regional Hospital (Other)
Responsible Party: Principal Investigator, Arne Astrup, professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: M198
Record Dates: First submitted 2010-06-08; First posted 2010-06-11 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Cardiovascular Diseases
Keywords: Apple; Apple pomace; Metabolomics; Gene expression; Lipid metabolism; Prevention; Antiinflammatory effect
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (No Intervention)
- Apples (Active Comparator)
  Interventions: Dietary Supplement: Apples
- Apple pomace (Active Comparator)
  Interventions: Dietary Supplement: Apple pomace

INTERVENTIONS:
Dietary Supplement: Apples — 550g of apples/day
  Arms: Apples
Dietary Supplement: Apple pomace — 22g apple pomace/day
  Arms: Apple pomace

SUMMARY:
The investigators will assess the protective and antiinflammatory effects of processed fruit and fruit fibre in overweight subjects with signs of metabolic syndrome. A single-blinded parallel study is conducted to investigate the protective effects of fruit fibre on colonic epithelium. Relevant signalling pathways related to cholesterol metabolism, vascular inflammation, oxidative defence, apoptosis and sterol metabolism will be targeted. Volunteers are randomly assigned one of three groups. They are instructed to follow a polyphenol and pectin restricted diet for six weeks. The last four weeks in this six week period, the restricted diet is supplemented with whole apples (550g/day), apple pomace (22g/day) or nothing. Blood, urine, faecal samples and colon biopsies are collected before and after the four weeks intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI over 30
* No daily medication
* Not strenuous exercise > 10hours/week
* No blood donation 3 months before or during the study

Exclusion Criteria:

* Smoking
* Simultaneous participation in other research projects
* Use of any dietary supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Blood lipid profile (triacylglycerol and total-, LDL- and HDL-cholesterol) | Measured at week 2
Blood lipid profile (triacylglycerol and total-, LDL- and HDL-cholesterol) | Measured at week 6

SECONDARY OUTCOMES:
Blood pressure | Measured at week 2
Blood pressure | Measured at week 6
Anthropometry (weight, height, waist and hip circumference) | Measured at week 2
Anthropometry (weight, height, waist and hip circumference) | Measured at week 6
Inflammatory marker (hs-CRP) | Measured at week 2
Inflammatory marker (hs-CRP) | Measured at week 6
Faeces analyses (metabolomics, pH, bile acids, short-chain fatty acids) | Measured at week 2
Faeces analyses (metabolomics, pH, bile acids, short-chain fatty acids) | Measured at week 6
Urine analyses (metabolomics) | Measured at week 2
Urine analyses (metabolomics) | Measured at week 6
Serum insulin, IGF-1 and IGFBP-3 levels | Measured at week 2
Serum insulin, IGF-1 and IGFBP-3 levels | Measured at week 6
Gene expression in white blood cells and colon tissue | Measured at week 2
Gene expression in white blood cells and colon tissue | Measured at week 6
Enzyme activity in lysed erythrocytes (glutathione peroxidase) | Measured at week 2
Enzyme activity in lysed erythrocytes (glutathione peroxidase) | Measured at week 6

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Bügel, PhD, Study Director — Department of Human Nutrition, LIFE, University of Copenhagen, Denmark
Locations (1):
- Department of Human Nutrition, LIFE, University of Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Yes